CLINICAL TRIAL: NCT03815851
Title: Relationship Between Prophylactic Drainage and Postoperative Complications (PPOI et al) in Crohn's Patients After Surgery
Brief Title: Relationship Between Prophylactic Drainage and Postoperative Complications (PPOI) in Crohn's Patients After Surgery
Acronym: RBPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, the ethics committee of the hospital, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: jinlingH201608
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial
Masking Description: Investigators, surgical team and patients were not blinded to the assignment. In the the drain group, a 28 G latex tube was placed in the pelvic cavity intraoperatively and in the no-drain group, no drain was positioned. 30-day postoperative complications were assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain group (Other): Place prophylactic drainage after surgery.
  Interventions: Device: prophylactic drainage
- No-drain group (Other): Not place prophylactic drainage after surgery.
  Interventions: Device: no prophylactic drainage

INTERVENTIONS:
Device: prophylactic drainage — place prophylactic drainage after surgery
  Arms: Drain group
Device: no prophylactic drainage — Not place prophylactic drainage after surgery
  Arms: No-drain group

SUMMARY:
For patients with Crohn's diseases，whether prophylactic abdominal drainage is necessary need further exploration. the present study is focusing on the necessity of prophylactic abdominal drainage in CD patients after surgery.

DETAILED DESCRIPTION:
In the past decades, surgical dogma meant the correct placement of a prophylactic drain, with the aim of reducing the incidence of anastomotic leakage, decreasing the needs of reoperation and avoiding potential postoperative ascites. However, recent randomized controlled trials (RCTs) and meta-analyses have suggested that prophylactic peritoneal drains have no benefits on postoperative outcomes.

Crohn's disease (CD), which is definitely different from CRC, is a chronic inflammatory disease with unknown pathogenesis. CD itself was the independent risk factor of multiple postoperative complications, including anastomotic leakage, intraperitoneal abscess and catheter-associated bloodstream infection.

In the present RCT, we hypothesize that non-prophylactic peritoneal drainage is associated with increased incidence of postoperative non-septic complications.

ELIGIBILITY:
Inclusion Criteria:

* Stricturing CD patients with American Society of Anesthesiologists (ASA) score of 1 to 2 undergoing elective small bowel or ileocecal resection and anastomosis.

Exclusion Criteria:

* Coexisting penetrating disease (fistula, abscess or phlegmona), enterostomy, strictureplasty only, short bowel (less than 150 cm), preoperative hypokalemia, diabetes or hyperglycemia (fasting plasma glucose >126 mg/dL), as well as chronic systemic disease of cardiovascular, respiratory et al.
* Patients who received ≥20 mg/d prednisolone or equivalent for over 6 weeks within 4 weeks before surgery; patients who received steroids, biologics or gastrointestinal motility drugs within 4 w prior to surgery; patients who remained on steroids within 1 day before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of prolonged postoperative ileus | postoperative 30 days
  incidence of prolonged postoperative ileus

SECONDARY OUTCOMES:
recurrence | postoperative 30 days and 1 year after surgery for endoscopic recurrence.
  time to first passage of flatus and stool, pain relief, postoperative length of stay (LOS), postoperative complications (defined as Clavien-Dindo) within 30 days after surgery, incisional SSIs, readmission rates, medical costs,blood markers,endoscopic recurrence at the anastomosis.

CONTACTS AND LOCATIONS:
Overall Officials: weiming zhu, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China